CLINICAL TRIAL: NCT05191940
Title: Phase II Trial of Hypo-fractionated Highly Conformal Radiotherapy for Locally Advanced Pancreatic Carcinomas
Brief Title: Radiotherapy for Locally Advanced Pancreatic Carcinomas (Phase II Trial)
Acronym: LAPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EBG MedAustron GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LAPC-MA-092021
Record Dates: First submitted 2021-12-16; First posted 2022-01-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Pancreas Cancer
Keywords: Particle Radiotherapy; Hypofractionated radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Particle radiotherapy (Other): According to the radiation plan using protons or carbon ions (between 25 and a maximum of 40 Gy). Planning Target Volume 1 : 25 Gy (Relative Biological Effectiveness) in 5 fractions of 5 Gy (Relative Biological Effectiveness) Planning Target Volume 2 : A simultaneous integrated boost (SIB) will be delivered to the Planning Target Volume 2: 40 Gy (Relative Biological Effectiveness) in 5 fractions of 8 Gy (Relative Biological Effectiveness).
  Interventions: Radiation: Particle-therapy using protons or carbon ions; Diagnostic Test: Blood sampling; Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Computertomography; Diagnostic Test: 18-F-FluorDesoxyGlukose Positron Emission Tomography-Computer Tomography (18F-FDG-PET-CT)

INTERVENTIONS:
Radiation: Particle-therapy using protons or carbon ions — According to the radiation plan (between 25 and a maximum of 40 Gy). Planning Target Volume 1 : 25 Gy (Relative Biological Effectiveness) in 5 fractions of 5 Gy (Relative Biological Effectiveness) Planning Target Volume 2 : A simultaneous integrated boost (SIB) will be delivered to the Planning Target Volume 2: 40 Gy (Relative Biological Effectiveness) in 5 fractions of 8 Gy (Relative Biological Effectiveness).
Diagnostic Test: Blood sampling — Evaluation before treatment-start, after treatment and follow-up period.
Diagnostic Test: Magnetic resonance imaging — For treatment planning as well as for follow-up radiological tumor assessment.
Diagnostic Test: Computertomography — For treatment planning as well as for follow-up radiological tumor assessment.
Diagnostic Test: 18-F-FluorDesoxyGlukose Positron Emission Tomography-Computer Tomography (18F-FDG-PET-CT) — For treatment planning as well as for follow-up radiological tumor assessment.

SUMMARY:
This is an interventional, single-arm, open-label study with high dose short course radiotherapy for patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is an interventional, open label, trial of definitive hypofractionated radiotherapy for patients with locally advanced pancreatic cancer.

Within this study radiotherapy shall be delivered with active scanning particle-therapy using proton- or carbon ions radiotherapy.

Particle therapy will be performed with a simultaneous integrated boost (SIB) treating a larger target volume, including elective lymph node stations and neural plexus, at a lower dose and boosting macroscopic disease.

The investigator will explore the efficacy of these treatment in a real world scenario in which patients are allowed to receive standard systemic treatment and standard surgical treatment (if conversion to resectability is achieved).

However, and in order to record and to gain better understanding of the influence of systemic therapies on the outcomes parameters of this study, patients will be sub-stratified in 3 groups: i) patients receiving FOLFIRINOX, ii) patients receiving Gemcitabine + Nanoparticle Albumin Bound Paclitaxel (NAB-Paclitaxel), iii) patients receiving other systemic therapies or not receiving antineoplastic systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has histologically or cytological confirmed diagnosis of pancreatic cancer (cases with radiological findings suspicious of pancreatic cancer AND elevated CA 19-9 may be enrolled even without positive cytology)
2. The patient is not candidate for radical surgical resection because of one or more of the following reasons:

   1. the patient is staged as locally advanced and with unresectable disease according to the international consensus definition. Specific criteria are: there is involvement of portal vein/superior mesenteric vein with bilateral narrowing/occlusion, exceeding the inferior border of the duodenum; or tumor contact/invasion of 180 or more degree of the superior mesenteric artery or of the truncus coeliacus; or tumor contact/invasion of the proper hepatic artery/ celiac artery; or tumor contact or invasion of the aorta.
   2. the patient is not a candidate for radical surgery because of radiographic or biochemical (CA 19-9) progression during neoadjuvant chemotherapy despite being initially classified as resectable or borderline resectable according to the international consensus definition.
   3. the patient is not candidate for radical surgery because of cN+ stage
3. The patient is not candidate to (further) neoadjuvant chemotherapy because of one or more of the following reasons:

   1. the patient is not fit for chemotherapy
   2. the patient has progressed under chemotherapy
   3. the patient has received neoadjuvant chemotherapy but is judged still not a candidate for explorative surgery.
4. Negative staging for distant metastasis
5. Age > 18 years
6. Karnofsky index ≥ 70
7. No tumor infiltration of stomach or duodenum
8. The patient is informed of the diagnosis and is able to give informed consent (Ability of patient to understand character and individual consequences of the study protocol)
9. Women of fertile age must have adequate conception prevention measures and must not breast feed
10. Signed Informed Consent (must be available before study inclusion)

Exclusion Criteria:

1. Non-exocrine tumors
2. Major medical or psychiatric comorbidities that contraindicate radiotherapy
3. Presence of distant metastasis
4. Pregnancy or unwilling to do adequate conception prevention
5. Lactating and unwilling to discontinue lactation
6. Men of procreative potential not willing to use effective means of contraception
7. Metallic prosthesis or other conditions - IF it prevents an adequate imaging for target volume definition or treatment planning at the discretion of the treating institution contraindicate radiotherapy e.g. active infections in the area
8. Previous abdominal radiotherapy
9. Severe hepatic or renal impairment at discretion of treating institution
10. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Locoregional tumor control | At two year
  Rate of locoregional tumor control at two year will be evaluated radiologically.
  This endpoint will be measured with the actuarial approach.

SECONDARY OUTCOMES:
Loco-regional progression-free survival | 104 weeks after therapy
  This endpoint will be measured with the actuarial approach. It will be assessed as the union of locoregional control and survival. Patient with loco regional recurrence will be considered failures. Deceased patient will also be considered failures. Patient lost to follow-up without evidence of locoregional recurrence will be censored. Distant metastasis and peritoneal carcinosis will be irrelevant respect to this endpoint.
Overall survival | Maximal 109 weeks
  This endpoint will be measured with the actuarial approach. All deaths will be considered failures, patient lost to follow-up will be censored.
Incidence of CTCAE v5.0 G4-5 toxicity | From enrollment to six months after radiation therapy initiation
  This endpoint will be scored as gross rate. The investigator will measure the number of patients experiencing at least one toxicity >= Grade 4 and >= Grade 5 and the number of events >= Grade 4 and >= Grade 5. The crude number will be divided by the total number of patients treated.
Patient reported Health-related Quality of Life, measured with Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) | Maximal 109 weeks
  Quality of life will be measured with Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) before radiation therapy and at each follow-up. The FACT-Hep has 27 (+ a subscale with 18 additional) questions, each of which is answered using a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Questions are phrased so that higher numbers indicate a better health state, leading to some items being reverse-scored. Questions measure the respondents' health state over the last 7 days in four subscales: Physical Well-Being (7 questions), Social/Family Well-Being (7 questions), Emotional Well-Being (6 questions), and Functional Well-being (7 questions). This disease-specific version of the FACT-Hep contain these four core subscales, with additional (18) questions appended to address disease-specific factors.
  The higher the score the better the Quality of Life.
Patient reported Health-related Quality of Life, measured with European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire-C30 | Maximal 109 weeks
  Quality of life will be measured with EORTC Quality of Life Questionnaire-C30 before radiation therapy and at each follow-up.
  Questionnaire developed to assess the quality of life of cancer patients. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / quality of life (QoL) represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Patient reported Health-related Quality of Life, measured with Brief Pain Inventory | Maximal 109 weeks
  Quality of life will be measured with Brief Pain Inventory before radiation therapy and at each follow-up.
  The Brief Pain Inventory (BPI) is a measurement tool for assessing clinical pain.The interference items were now presented with 0-10 scales, with 0=no interference and 10=interferes completely.
Incidence of CTCAE v5.0 Grade 2 - Grade 5 acute, subacute and late toxicities | 104 weeks after therapy
  The number of events, their grade and their time course will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Fossati, M.D., Principal Investigator — EBG MedAustron GmbH
Locations (1):
- EBG MedAustron GmbH, Wiener Neustadt, Lower Austria, Austria